CLINICAL TRIAL: NCT02455011
Title: A Randomized, Placebo-controlled, Double-blind, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Single and Repeated Subcutaneous (SC) Doses of REMD-477 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of REMD-477 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R477-201
Record Dates: First submitted 2015-05-20; First posted 2015-05-27 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — volagidemab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- REMD-477 Treatment A (Experimental): Administered as a single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477
- Matching placebo (Placebo Comparator): Placebo administered as single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477
- REMD-477 Treatment B (Experimental): Administered as a single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477
- REMD-477 Treatment C (Experimental): Administered as a single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477
- REMD-477 Treatment D (Experimental): Administered as a single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477
- REMD-477 Treatment E (Experimental): Administered as a single and repeated SC doses in subjects with Type 2 Diabetes
  Interventions: Biological: REMD-477

INTERVENTIONS:
Biological: REMD-477

SUMMARY:
This is a randomized, placebo-controlled, double-blind, dose escalation study to evaluate safety, tolerability, PK and PD of single and repeated SC doses of REMD-477 in Type 2 diabetic subjects. The study will be conducted at multiple sites in the United States and will enroll approximately 102 subjects with Type 2 diabetes who are either treatment-naïve, controlled with diet and exercise or treated with oral antidiabetic medications.

DETAILED DESCRIPTION:
The study will consist of three parts: Part A - Dose Escalation, Part B - Adaptive Dose Cohort, and Part C - REMD-477 in Combination with Metformin. Part A includes 5 cohorts that will be enrolled and dosed sequentially at escalating doses. Each cohort will consist of 12 subjects randomized in a 3:1 (active: placebo) fashion. Part B includes a single dose cohort that will enroll 12 subjects (9 on active treatment and 3 on placebo) with dose level and frequency determined by a Dose Level Review Meeting (DLRM)Committee. Part C includes 2 cohorts of T2DM patients currently treated with metformin alone, and each cohort will consist of 15 subjects (10 on active treatment and 3 on placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years old, inclusive, at the time of screening;
* Females of non-child bearing potential must be ≥1 year post-menopausal (confirmed by a serum follicle-stimulating hormone (FSH) levels ≥ 40 IU/mL) or documented as being surgically sterile, and females of child bearing potential must use two medically acceptable methods of contraception;
* Male subjects must be willing to use clinically acceptable contraception during treatment and for 2 months after the last administration of REMD-477;
* Normal or clinically-acceptable physical examination, laboratory test values, and 12-lead ECG (reporting heart rate and PR, QRS, QT, and QTcF) at screening;
* Body mass index between 23 and 40 kg/m2, inclusive, at screening;
* Diagnosed with Type 2 diabetes as defined by the current American Diabetes Association (ADA) criteria;
* Subjects in Parts A and B only: Treatment-naive, controlled with diet and exercise, or treated with oral antidiabetic medications and willing to wash-out and discontinue oral medications during the study;
* Fasting plasma glucose 126 - 270 mg/dL (7-15 mM), inclusive, at screening and at re-test on Day -1;
* Subjects in Parts A and B only: Screening HbA1c of 7.0-10 % inclusive for subjects not currently taking any oral antidiabetic medications, or 6.5-9.5% for subjects receiving acceptable oral antidiabetic medications;
* Subjects in Part C only: Screening HbA1c of 7.5-10 % inclusive for subjects on stable doses of metformin.

Exclusion Criteria:

* History of drug or alcohol abuse within the last 6 months or a positive illegal drug urine test result;
* History or family history of pancreatic neuroendocrine tumors or multiple endocrine neoplasia;
* History or family history of pheochromocytoma;
* Known or suspected susceptibility to infectious disease (eg, taking immunosuppressive agents or has a documented inherited or acquired immunodeficiency);
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C antibodies (HepC Ab);
* Participation in an investigational drug or device trial within 30 days of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known, whichever period is longer;
* Blood donor, or blood loss>300 mL, within 30 days of Day 1;
* Recent use (6 weeks prior to Screening) of thiazolidinediones, >half-maximal dose sulfonylurea agent therapy, or any injectable antidiabetic agents (exenatide and other injectable GLP-1 agonists, insulin and insulin analogs, etc.);
* Other gastrointestinal, cardiac, renal and CNS (i.e. hypoglycemia unawareness) conditions specific to diabetes that would pose additional risk to subject's safety or interfere with the study evaluation, procedures or completion;
* Lipid panel profiles of non-HDL-C (total cholesterol minus HDL-C) >219 mg/dL, LDL-C >189 mg/dL, and/or fasting triglycerides >499 mg/dL;
* Female subject is pregnant or breastfeeding.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events per subject, including changes in vital signs, physical and neurological examinations, laboratory safety tests and ECGs | 141 Days

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile (parameters including maximum observed concentration (Cmax), area under the curve (AUC) serum-concentration, clearance, and half-life (t1/2) after single and repeated SC doses. | 141 Days
Changes in fasting glucose and insulin levels following single and repeated SC doses of REMD-477. | 141 Days
Changes in glucose and insulin AUC following a Mixed Meal Tolerance Test. | Day 29, Day 57 and Day 85
Incidence of REMD-477 neutralizing and non-neutralizing antibodies | 141 Days
Incidence of elevated alanine transaminase (ALT) or aspartate transaminase (AST) values >3x the upper limit of normal with concomitant >2x increases in alkaline phosphatase (ALP) and/or >2x total bilirubin. | 141 Days
Incidence and severity of elevated amylase and lipase values at >2.5x ULN after study treatment | 141 Days
Geometric mean ratio to baseline over time of AST, ALT, ALP and total bilirubin. | 141

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami, Florida
  - San Antonio, Texas
  - Renton, Washington